CLINICAL TRIAL: NCT04568473
Title: Effectiveness of Bioactive Resin Based Varnish and Fluoride Varnish Containing Xylitol-coated Particles Versus Sodium Fluoride Varnish in Management of Teeth Hypersensitivity in Adult Patients Over Eight Weeks: a Randomized Clinical Trial.
Brief Title: Effectiveness of Bioactive Resin Varnish and Fluoride Containing Xylitol Varnish in Management of Teeth Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Abd El-Fattah, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU-HAElFattah
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2020-09

CONDITIONS: Tooth Hypersensitivity
Keywords: Hypersensitivity; Sodium Fluoride; Xylitol coated Calcium and Phosphate; BioSmart Light Cured Protective Shield
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity | interventions — PRG Barrier Coat

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PRG Barrier Coat (SHOFU Inc., Japan) (Experimental): BioSmart Light Cured Protective Shield with bioactive S-PRG (Surface Pre-Reacted Glass ionomer) filler technology.
  S-PRG filler possesses a three-layer structure with a stabilized glass-ionomer-like structure surrounding multifunctional glass fillers, and is subsequently protected by a surface modified layer.
  Interventions: Other: EMBRACE™ Varnish by (Pulpdent Corporation, USA)
- EMBRACE™ Varnish (Pulpdent Corporation, USA) (Experimental): Resin-based 5% sodium fluoride with CXP™ (Xylitol-coated Calcium and Phosphate) technology for unsurpassed fluoride release.
  The incorporation of CXP™ (xylitol-coated calcium and phosphate) in a permeable resin matrix that does not separate, purportedly drives the sustained, time-released properties of this varnish
  Interventions: Other: PRG Barrier Coat (By SHOFU Inc., Japan)
- Duraphat® (Colgate Palmolive Company, New York, NY) (Active Comparator): It is attributed to the reactivity of the fluoride by adsorbing to the surface and attracting calcium ions forming loosely-bound calcium fluoride (CaF2)- like reservoir which is also considered responsible for the anticaries mechanism and protection against cariogenic acid attack.
  Interventions: Other: PRG Barrier Coat (By SHOFU Inc., Japan); Other: EMBRACE™ Varnish by (Pulpdent Corporation, USA)

INTERVENTIONS:
Other: PRG Barrier Coat (By SHOFU Inc., Japan) — PRG Barrier Coat (By SHOFU Inc., Japan) is a bioactive, resin-based varnish based on the proprietary Giomer concept which incorporates the patented bioactive S-PRG (Surface Pre-Reacted Glass ionomer) filler technology, where a unique combination of six beneficial ions are actively gradually released to provide a smart solution to revolutionize dentin hypersensitivity protocol
  Other Names: Bio-smart Light Cured Protective Shield with bioactive S-PRG (Surface Pre-Reacted Glass ionomer)
  Arms: Duraphat® (Colgate Palmolive Company, New York, NY); EMBRACE™ Varnish (Pulpdent Corporation, USA)
Other: EMBRACE™ Varnish by (Pulpdent Corporation, USA) — 5% sodium fluoride with CXP™ (Xylitol-coated Calcium and Phosphate) technology for unsurpassed fluoride release and it is considered as a novel method of delivering remineralizing ions (Calcium and Phosphate) in combination with xylitol. The incorporation of CXP™ in a permeable resin matrix that does not separate, purportedly drives the sustained, time-released properties of this varnish.it has ten times more fluoride release over a 4-hour period than the leading varnish brand, in addition, it also releases bioavailable calcium and phosphate ions which are nano-coated with xylitol.
  Arms: Duraphat® (Colgate Palmolive Company, New York, NY); PRG Barrier Coat (SHOFU Inc., Japan)

SUMMARY:
Will the use of Bio-smart Light Cured Protective Shield with bioactive S-PRG filler or the use of Sodium Fluoride with Xylitol-coated Calcium and Phosphate (CXP™) Varnish be able to reduce the teeth hypersensitivity similar to Sodium Fluoride Varnish?

DETAILED DESCRIPTION:
The null hypothesis tested in this study, that there is no difference in clinical effectiveness between bio-smart Shield with bioactive S-PRG filler and Fluoride varnish containing Xylitol-coated Calcium and Phosphate (CXP™) Compared to Sodium Fluoride Varnish in management of hypersensitivity in adult patients after 3 minutes, 2, 4 and 8 weeks.

P (Population): Patient with Teeth Hypersensitivity.

Intervention-1: Bio-smart Light Cured Protective Shield with bioactive S-PRG (Surface Pre-Reacted Glass ionomer) filler technology (PRG Barrier Coat) by (By SHOFU Inc., Japan).

Intervention-2: 5% Sodium Fluoride with Xylitol-coated Calcium and Phosphate (CXP™) Varnish (Embrace™ Varnish) by (Pulpdent Corporation)

C (Comparator): 5% Sodium Fluoride Varnish (Duraphat®) by (Colgate Palmolive Company, New York, NY)

O (Outcome):

* Primary Outcome: Pain due to Hypersensitivity
* Secondary Outcome: Dentinal tubules occlusion

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of hypersensitive areas on facial surfaces of the teeth (incisors, cuspids, bicuspids, and first molars with exposed cervical dentin)

  * Teeth scoring pain (VAS score: greater than or equal to 5) during application of stimulus (air blast, thermal and tactile sensitivity test).
  * Patients with good oral hygiene.
  * Co-operative patients who show interest to participate in the study accept the 2-months follow-up period.

Exclusion Criteria:

* Patients participating in another dental study that may alter the results of this study.
* A medical condition that could hinder the accuracy of pain reporting (e.g., pain disorders).
* Any chronic medical condition that requires the regular use of anti-inflammatory pain medications.
* Patients used or applied a desensitizing varnish within the last four weeks.
* Patients with dental problems; chipped teeth, defective restorations, fractured Un-displaced cuspids or deep dental caries.
* Patients with orthodontic appliances, or bridge work that might interfere with evaluation
* Lack of patient's approval and compliance.
* Patients who are allergic to any ingredients will be used in the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Amount of pain due to dentin hypersensitivity (evaporative stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | Baseline
  Amount of Pain arising from dentin hypersensitivity in non-carious cervical lesions stimulated by air blast measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (evaporative stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 3 minutes
  Amount of Pain arising from dentin hypersensitivity in non-carious cervical lesions stimulated by air blast measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (evaporative stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 2 weeks
  Pain arising from dentin hypersensitivity in non-carious cervical lesions stimulated by air blast measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (evaporative stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 4 weeks
  Pain arising from dentin hypersensitivity in non-carious cervical lesions stimulated by air blast measured by a 10 cm Visual Analogue Scale (from 0 to 10) . Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (evaporative stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 8 weeks
  Pain arising from dentin hypersensitivity in non-carious cervical lesions stimulated by air blast measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort

SECONDARY OUTCOMES:
Amount of pain due to dentin hypersensitivity (Thermal stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | Baseline
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (Thermal stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 3 minutes
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (Thermal stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 2 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (Thermal stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 4 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (Thermal stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 8 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by cold water measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (Tactile stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | Baseline
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (Tactile stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 3 minutes
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (Tactile stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 2 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (Tactile stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 4 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Amount of pain due to dentin hypersensitivity (Tactile stimulus) using Visual Analogue Scale, (0) indicates No Pain and (10) indicates maximum Pain | 8 weeks
  Pain arising from dentin hypersensitivity in non-carious lesions stimulated by tactile stimulation with a probe measured by a 10 cm Visual Analogue Scale (from 0 to 10). Dentin hypersensitivity will be measured, with the score of zero being a pain-free response and score of 10 being excruciating pain or discomfort
Dentinal Tubule Occlusion | Baseline
  Scanning Electron Microscope and digital image analysis measuring the surface area of patent dentinal tubules
Dentinal Tubule Occlusion | 8 weeks
  Scanning Electron Microscope and digital image analysis measuring the surface area of patent dentinal tubules

CONTACTS AND LOCATIONS:
Overall Officials: Heba AE Mohamed, Master's, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
The personal data of the participants will not present on the protocol form and it would be maintained secured for 10 years after the trial for protection of participants' privacy and civil rights.

REFERENCES:
- [Derived] Abd El-Fattah Mohamed H, Ezzeldin Mohamed D, Hassanein E, Salah El-Din Hamza HE. In vivo and in situ evaluation of innovative approaches in dentin hypersensitivity treatment. BMC Oral Health. 2025 Apr 18;25(1):593. doi: 10.1186/s12903-025-05865-y. PMID 40251520